CLINICAL TRIAL: NCT01917292
Title: Periodontal Intervention Improves Vascular Function Among Chinese Prehypertensive Adults With Periodontitis
Brief Title: Impact of Periodontal Intervention on Vascular Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Junying Yang, professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20130718emp; 31270992 (Registry Identifier: National Natural Science Foundation of China)
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Periodontitis; Prehypertension
Keywords: Periodontitis; Prehypertension; Periodontal Intervention
MeSH Terms: conditions — Chronic Periodontitis; Prehypertension; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Periodontal care (Other)
  Interventions: Procedure: Periodontal care
- One-Stage Full-Mouth Disinfection (Experimental)
  Interventions: Procedure: One-Stage Full-Mouth Disinfection

INTERVENTIONS:
Procedure: One-Stage Full-Mouth Disinfection — 1. Basic oral hygiene instructions
  2. Dental extractions will be performed (only in cases of teeth that could not be saved)
  3. Standard cycle of supragingival ultrasonic scaling and polishing
  4. Scaling and root planning after the administration of local anesthesia, four quadrants in one session
  5. Minocycline Hydrochloride Ointment (Periocline, OraPharma) were delivered locally into the periodontal pockets
  Arms: One-Stage Full-Mouth Disinfection
Procedure: Periodontal care — 1. Basic oral hygiene instructions
  2. Standard cycle of supragingival ultrasonic scaling and polishing
  Arms: Periodontal care

SUMMARY:
The purpose of this study is to determine the effect of periodontal intervention on vascular dysfunction among Chinese prehypertensive adults with moderate to severe periodontal disease.

DETAILED DESCRIPTION:
Periodontitis is one of the low-grade chronic diseases, and it is the principal cause of tooth loss among middle-aged and elderly. Recently, epidemiological data indicate that patients with periodontitis are associated with increases in blood pressure levels and hypertension prevalence. Furthermore, studies from cross-sectional investigations demonstrate that hypertensive patients with periodontitis may enhance the risk and degree of vascular damage. Therefore, periodontal therapy is a novel therapeutic strategy to prevent the occurrence of BP elevation and retard the development vascular injury.

The term "prehypertension" indicates those with BPs ranging from 120 to 139 mm Hg systolic and/or 80 to 89 mm Hg diastolic blood pressure. Accumulating evidence suggests that subjects with prehypertension is associated with higher incidence of atherosclerotic vascular disease. However, until now there are no available data to investigate the influence of periodontitis on prehypertension and whether periodontal intervention may reduce the BP rise in subjects with prehypertension and improve the vascular function. We hypothesized that periodontitis leads to elevation in BP and periodontal therapy improves vascular function in subjects with prehypertension. To address these assumptions, The present study is designed to study the effect of periodontal intervention on blood pressure and vascular function and inflammatory biomarkers among Chinese prehypertensive adults with moderate to severe periodontal disease, and determine whether intensive periodontal therapy improves these measures over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older
2. Moderate to severe generalized periodontitis(probing pocket depths of >6 mm and Marginal alveolar bone loss of >30%) with 50% or more of their teeth affected
3. Have at least 16 natural teeth excluding third molars
4. BPs ranging from 120 to 139 mm Hg systolic and/or 80 to 89 mm Hg diastolic blood pressure
5. Provide informed consent and willingness to cooperate with the study protocol

Exclusion Criteria:

1. History of antibiotic use in the previous three months
2. Pregnant or lactating females
3. Systemic diseases such as diabetes, HIV/AIDS, liver disease, chronic renal failure, tuberculosis, and autoimmune diseases
4. Medical history of cardiovascular disease: Acute myocardial infarct, stable angina, unstable angina, heart failure, atrial fibrillation, atrioventricular blockade, peripheral vascular disease, cerebrovascular accident, hypertension
5. Patients who received periodontal treatment within the last 6 months
6. Patients who require antibiotic prophylaxis before examination or treatment
7. Patients with mental retardation and dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Number of Endothelial Microparticle at 6 months | Baseline; 1 month post periodontal therapy; 3 months post periodontal therapy; 6 months post periodontal therapy
Change from Baseline in the Blood Pressure at 6 months | Baseline; 1 month post periodontal therapy; 3 months post periodontal therapy; 6 months post periodontal therapy

SECONDARY OUTCOMES:
Change in Brachia-ankle Pulse Wave Velocity(baPWV) | Baseline; 1 month post periodontal therapy; 3 months post periodontal therapy; 6 months post periodontal therapy
Changes in high-sensitivity C-Reactive Protein(hs-CRP) and Interleukin-6(IL-6) | Baseline; 1 month post periodontal therapy; 3 months post periodontal therapy; 6 months post periodontal therapy
  Compare the changes of traditional inflammatory biomarkers：hs-CRP and IL-6 over a 6-month follow-up period.
Expression of the Long non-protein-coding RNA(lncRNA) and microRNA | baseline
Changes in Malondialdehyde(MDA) and Superoxide Dismutase(SOD) | Baseline; 1 month post periodontal therapy; 3 months post periodontal therapy; 6 months post periodontal therapy
Change in Periodontal Inflamed Surface Area(PISA) | Baseline; 3 months post periodontal therapy; 6 months post periodontal therapy
  Bleeding on probing(BOP), clinical attachment loss (CAL) and gingival recession(GR) are measured to calculate the PISA.The PISA reflects the surface area of bleeding pocket epithelium in square millimetres.
Change in Endothelium-dependent Brachial Artery Flow-mediated Dilation(FMD) | Baseline; 1 month post periodontal therapy; 3 months post periodontal therapy; 6 months post periodontal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ying Yang, Master, Study Director — First Affiliated Hospital, Sun Yat-Sen University; Jun Tao, M.D.,phD., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhou QB, Xia WH, Ren J, Yu BB, Tong XZ, Chen YB, Chen S, Feng L, Dai J, Tao J, Yang JY. Effect of Intensive Periodontal Therapy on Blood Pressure and Endothelial Microparticles in Patients With Prehypertension and Periodontitis: A Randomized Controlled Trial. J Periodontol. 2017 Aug;88(8):711-722. doi: 10.1902/jop.2017.160447. Epub 2017 Apr 28. PMID 28452620